CLINICAL TRIAL: NCT07089511
Title: Cord Blood Platelet Poor Plasma Eye Drops
Acronym: CB3P-ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CB3P-ED; PNRR-MCNT2-2023-12377596 (Other Grant/Funding Number: Ministero della salute)
Record Dates: First submitted 2025-07-16; First posted 2025-07-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-07

CONDITIONS: Dry Eye
Keywords: Cord Blood Platelet Poor Plasma; dry eye disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CB3P-ED (Experimental)
  Interventions: Other: CB3P-ED + 0.1% cyclosporine eye drops
- 0.15% hyaluronic acid (Active Comparator)
  Interventions: Other: 0.15% hyaluronic acid + 0.1% cyclosporine eye drops

INTERVENTIONS:
Other: CB3P-ED + 0.1% cyclosporine eye drops — Combination of CB3P-ED + 0.1% cyclosporine eye drops
  Arms: CB3P-ED
Other: 0.15% hyaluronic acid + 0.1% cyclosporine eye drops — Combination of 0.15% hyaluronic acid + 0.1% cyclosporine eye drops
  Arms: 0.15% hyaluronic acid

SUMMARY:
Dry eye disease (DED) is a prevalent ocular condition characterized by the disruption of the ocular surface's homeostasis. It affects a significant portion of the population, particularly women and older individuals. The impact of DED on the healthcare system and patients' quality of life is substantial, with approximately 30 million adult patients (14.5%) reporting DED symptoms in the US. Global mapping studies have shown that DED prevalence ranges from 5% to 50% of the population. While chronic instillation of artificial tears is the main treatment strategy for DED, it is often ineffective in moderate to severe cases associated with corneal inflammation.

Innovative therapeutic approaches using human serum and platelet derivatives have shown promising results in tear substitution. Umbilical cord blood plasma, which contains natural tissue regenerative and immunomodulatory factors, has demonstrated positive effects on corneal epithelial cells and clinical efficacy in observational studies. This study aims to develop a randomized clinical trial protocol to compare the clinical efficacy of artificial tears (control arm) and human platelet poor plasma from umbilical cord blood (treatment arm) in the treatment of DED.

The results of this clinical trial will contribute to understanding the clinical efficacy of umbilical cord blood plasma eye drops compared to artificial tears in the treatment of moderate to severe DED.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years.
2. Male or female.
3. Diagnosis of Dry Eye Disease (DED) with severe keratitis and ocular discomfort related to DED, defined as follows:

   Corneal Fluorescein Staining (CFS) score of 3, 4, or 5 on the modified Oxford scale in at least one eye at the Baseline Visit, combined with at least one of the following criteria:

   i. Schirmer test without anesthesia with a score <10 mm/5 min in the same eye at the Baseline Visit.

   ii. Ocular Surface Disease Index (OSDI) score of at least 30, or presence of at least two moderate to severe dry eye symptoms with a severity score above 50 (severity assessed on a scale of 0 to 100), including any of the following symptoms: burning/stinging, foreign body sensation, ocular dryness, ocular pain, and blurred/decreased vision at the Baseline Visit.
4. Ability to understand and comply with the protocol requirements (as judged by the investigator).
5. Provision of written informed consent and privacy authorization prior to initiation of any study procedures.
6. At least 3 months of conventional treatment use (cyclosporine 1 mg/ml and/or hyaluronic acid) for DED prior to the Baseline Visit.
7. Willingness and ability to undergo all scheduled examinations and visits during the study.

Exclusion Criteria

1. Active herpetic keratitis or history of ocular herpes.
2. History of ocular trauma or ocular infection (viral, bacterial, fungal, protozoal) within 90 days prior to the Baseline Visit.
3. Any ocular disease other than Dry Eye Disease (DED) requiring topical ocular treatment during the study period.
4. Ocular rosacea and/or severe blepharitis.
5. Progressive pterygium.
6. Concurrent ocular allergy (including seasonal conjunctivitis) or chronic conjunctivitis other than dry eye.
7. Planned insertion of temporary punctal plugs during the study period.
8. Best corrected visual acuity (BCVA) score ≤ 0.1 (decimal notation) in either eye.
9. Unstable systemic disease within 30 days prior to the Baseline Visit (e.g., diabetes with out-of-range blood glucose, thyroid dysfunction, uncontrolled autoimmune disease, ongoing systemic infections) or conditions judged by the investigator as incompatible with study participation.
10. Presence or history of severe systemic allergy.
11. Known hypersensitivity to any of the products used in the study (cyclosporine, fluorescein, lissamine green, hyaluronic acid) or their components.
12. History of ocular malignancy.
13. History of malignancy (other than ocular) within the last 5 years.
14. Any changes within 30 days prior to the Baseline Visit, or anticipated changes during the study, in the dosage of systemic medications that may affect dry eye condition [e.g., estrogen-progesterone or other estrogen derivatives, pilocarpine, isotretinoin, tetracycline, antihistamines, tricyclic antidepressants, anxiolytics, antimuscarinics, beta-blockers, phenothiazines, omega-3 fatty acids, systemic corticosteroids]. These treatments are permitted during the study provided their dosage remains stable throughout.
15. Any changes in systemic immunosuppressive therapy within 30 days prior to the Baseline Visit or anticipated changes during the study.
16. History of substance abuse or alcohol dependence.
17. Presence or history of any systemic or ocular disorder, condition, or disease that could interfere with the conduct of study procedures or interpretation of study results.
18. Pregnancy or breastfeeding at the time of the Baseline Visit.
19. Women of childbearing potential unwilling to use a highly effective method of contraception (see section 5.2.2) from the Baseline Visit throughout the treatment period and up to 2 weeks after study completion. Postmenopausal women (defined as ≥ 2 years without menstruation) are exempt from contraception requirements.
20. Participation in a clinical trial involving an investigational product within 30 days prior to the Baseline Visit.
21. Concurrent participation in another clinical trial during the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Corneal Fluorescein Staining | month 2
  The difference in the mean change from baseline in the corneal and conjunctival staining (CFS) score at the 2-month visit between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Viola, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No